CLINICAL TRIAL: NCT04748302
Title: Impaired Glucose Tolerance and Cognition in MS
Status: Terminated | Type: Observational
Why Stopped: COVID
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, J. Nicholas Brenton, MD, Principal Investigator, University of Virginia
Other Study IDs: 21791
Record Dates: First submitted 2019-09-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot study to compare cognitive performance in two groups of subjects with multiple sclerosis; those with normal glucose tolerance and those with impaired glucose tolerance. The study consists of a 2 hour oral glucose tolerance test, patient reported outcomes, a series of cognitive functioning tests, and outpatient physical assessment using a pedometer.

DETAILED DESCRIPTION:
Investigators plan to recruit 100 compliant patients with relapsing-remitting MS who are willing to come fasting for an oral glucose tolerance test to determine the relationship between glucose tolerance and cognition in MS patients.

Eligible study subjects expressing interest will be given a copy of the consent to review and will have the opportunity to ask questions. If the subject passes screening, they will be invited for their research visit. Signed consent form at the visit will be obtained before any study related procedures take place.

Baseline Measurements: Measurements for all subjects will include age, race/ethnicity, sex, weight, height, waist circumference, blood pressure. Relevant medical history, current medications, and family history diabetes will be reviewed and documented by both subject report and medical records. If the subject is a woman of child-bearing ability, urine pregnancy test will be done in order to exclude pregnant subjects. All subjects will then have an IV placed and have blood drawn to measure their fasting blood glucose level. Fasting blood glucose above 126 ug/dl would be a screen failure for this study.

Labs: The following labs will be drawn for all subjects.

* Blood glucose management (hemoglobin A1C, insulin-like growth factor, insulin) - these tests show how your body manages sugar
* Lipids & Metabolic Markers (fasting lipid profile, leptin, adiponectin) - these measure signal proteins in your blood for metabolism
* Cytokine profile - to assess impact of blood sugar and inflammatory factors (molecules that may indicate how well your immune system works) on recovery from your MS relapse
* Sodium level - to assess how your body uses water
* Vitamin D25 - measures amount of vitamin D in your body
* Neuro-filament light measurement - marker of neurodegeneration

Oral Glucose Tolerance Test: After baseline measurements and labs are obtained, subjects will drink a 75g glucose drink. Labs (blood glucose and insulin levels) will be drawn every 30 minutes for a total of 2 hours.

In between blood draws, the subjects will undergo functional testing and complete questionnaires. A neurological exam will also be done that includes 8 functional systems: pyramidal, cerebellar, sensory, brainstem, vision, bowel and bladder, mental, and ambulation.

Cognitive testing will include the single Digit Modalities Test (SDMT) which is a timed test measuring thinking speed associating numbers and symbols as well as the cogstate which is a computer based assessment that tests cognitive levels.In addition, all subjects will undergo the sloan Low Contrast Vision testing (LCVA) which assesses your ability to see letters at different contrast levels.

Subjects will complete questionnaires that will ask about their fatigue level, daily activities, sleep habits, and how they are feeling physically, emotionally, and mentally.

At the end of the visit subjects will be discharged to home with an ActiGraph GT3X+ accelerometer, a waist-worn device, to measure community-based ambulation (a measure of physical activity). Subjects will complete 7 days of wear-time and will return accelerometers by mail.

This study only requires one visit to the University of Virginia and will take approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Diagnosis of Clinically Isolated Syndrome (CIS) or Relapsing Remitting Multiple Sclerosis (RRMS) confirmed by McDonald 2010 criteria
* EDSS < 6.5 at time of visit

Exclusion Criteria:

* Diabetes type I or II
* use of glucose regulating medications
* fasting blood glucose of > 126 mg/dl
* known cardiac or respiratory disease
* morbid obesity (BMI >40)
* steroid exposure within 4 weeks of enrollment
* pregnancy or current use of hormone replacement therapy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Persons with RRMS or CIS between the ages of 18-59 who are not diabetic or on glucose regulating medications.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of glucose intolerance on clinical outcome measure of disability. | 1 year
  The expanded disability scale (EDSS) will be used to determine a subjects level of disability. This value will then be compared to the subjects category of glucose intolerance, measured by yes (abnormal glucose tolerance) or no (normal glucose tolerance). This is on a score from 0 (no disability) to 8 (bedridden)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States